CLINICAL TRIAL: NCT03508076
Title: Efficacy of Vibrating Capsule in Patients With Chronic Constipation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Deputy Director, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Vibrating Capsule
Record Dates: First submitted 2017-04-23; First posted 2018-04-25 (Actual); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Chronic Constipation
Keywords: Vibrating Capsule; Efficacy and Safety; Chronic Constipation; different vibrating modes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sham Capsule (Sham Comparator): Patients swallowed 1 sham Vibrating capsule with water every three days，recorded his defecation time, defecation frequency and bristol score.The total capsule need to take 12.
  Interventions: Device: Sham Capsule
- Vibration Capsule of low level (Experimental): Patients swallowed 1 low level vibration Capsule Vibrating capsule with water every three days，recorded his defecation time, defecation frequency and bristol score.The total capsule need to take 12.
  Interventions: Device: Vibrating Capsule
- Vibration Capsule of high level (Experimental): Patients swallowed 1 high level vibration Capsule Vibrating capsule with water every three days，recorded his defecation time, defecation frequency and bristol score.The total capsule need to take 12.
  Interventions: Device: Vibrating Capsule

INTERVENTIONS:
Device: Vibrating Capsule — Patients in this group would be treated with Vibrating Capsule
  Arms: Vibration Capsule of high level; Vibration Capsule of low level
Device: Sham Capsule — Capsules can't vibrate but look the same as Vibrating Capsule
  Arms: Sham Capsule

SUMMARY:
Constipated patients in the participating center from February 2017 to June 2018 (anticipated) were prospectively enrolled. Number of defecation per week，Bristol score，and Colon transmission experiment were compared with the constipated patients before treatment.

DETAILED DESCRIPTION:
Constipation affects the quality of life of patients, some patients abuse laxatives or repeated medical treatment, increased medical costs. At present, the main treatment of constipation is to adjust life style, medicine, psychotherapy, biofeedback and surgical treatment. However, the above methods are associated with adverse reactions, and the patient's satisfaction is still low. A new approach is needed to solve this clinical problem.

Investigators have developed a vibration capsule that can be adjusted in different modes.

Preliminary animal experiments showed that the capsule was safe and increased the number of defecation.

This study is a clinical research for patients with constipation, to explore the effect in different vibrating modes in patients with constipation and tract emptying transmission and its effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged form 18 to 80
* Clinical diagnosis of functional constipation
* Must be able to swallow vibrating capsule

Exclusion Criteria:

* complex history of gastrointestinal diverticula, obstruction, ulcer, bleeding, stenosis or fistula.
* recent use of banned drugs.
* patients who are preparing for mri.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
defecation frequency | 8 weeks
  the average weekly defecation frequency

SECONDARY OUTCOMES:
Bristol Stool Chart | 8 weeks
  Record the BSC of each defecation.
first defecation | 8 weeks
  The time of complete defecation after taking the capsule for the first time

CONTACTS AND LOCATIONS:
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
We may share IPD when we finish this research

REFERENCES:
- [Result] Yu J, Qian YY, He CH, Zhu SG, Zhao AJ, Zhu QQ, Shao CW, Wang TG, Wang Y, Ding GL, Liao Z, Li ZS. Safety and Efficacy of a New Smartphone-controlled Vibrating Capsule on Defecation in Beagles. Sci Rep. 2017 Jun 6;7(1):2841. doi: 10.1038/s41598-017-02844-4. PMID 28588191